CLINICAL TRIAL: NCT01108653
Title: A Structuralised Sick-leave Program Compared to Usual Care Sick Leave Management in Patients After an Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Other Government)
Responsible Party: Oslo University Hospital. Trondheimsveien 235,0514 Oslo, Norway.(Professor Stefan Agewall), Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REK sør-øst B:2009/719b
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-01

CONDITIONS: Myocardial Infarction
Keywords: Cardiovascular diseases; Heart diseases; Myocardial infarction; Rehabilitation; Health Economy; Randomized controlled trials; Non ST Elevation Myocardial Infarction (NSTEMI); Cost analysis; Sick-leave; Quality of Life
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases; Heart Diseases; Non-ST Elevated Myocardial Infarction

ARMS (2):
- Group 1: Usual care sick-leave management (Other)
  Interventions: Other: Usual care sick-leave management
- Group 2: Structuralised sick-leave program (Other)
  Interventions: Other: Structuralised sick-leave program

INTERVENTIONS:
Other: Usual care sick-leave management — Patients randomized to usual care. Follow up after discharge by general practitioner (GP) according to local practice.
  Arms: Group 1: Usual care sick-leave management
Other: Structuralised sick-leave program — Patients randomized to the structuralized program will get full time sick-leave for 2 weeks after discharge.Cardiologist will be responsible for individual adaption of each patient's sick-leave and follow-up.
  Arms: Group 2: Structuralised sick-leave program

SUMMARY:
In this study the investigators aim at comparing the effect on quality of life and the cost-effectiveness of a structuralised sick-leave program compared to usual care sick leave management in patients after an acute non ST myocardial infarction(NSTEMI).The investigators hypothesize that a structuralised sick-leave program after an acute NSTEMI is cost-effective without a negative effect on quality of life compared to usual care management in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute NSTEMI who are revascularized.
* 65 years old or less
* Self caring
* Adequately literate in Norwegian
* Have a regular work in at least 50% position.

Exclusion Criteria:

* Patients not willing to participate
* Professional drivers
* Patients with alcohol or drug abuse
* Severe complications after the myocardial infarction such as malignant arrythmias, heart failure and major bleedings.
* Patients with recent CABG ( coronary artery bypass graft operation) within the last 6 months.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Cost effectiveness | one year
  In order to evaluate resource use (costs) all patients will be asked to fill in a questionnaire at baseline and after 6 and 12 months. Total costs and mean costs will be calculated in the two different follow-up modalities.

SECONDARY OUTCOMES:
Quality of Life measures are estimated at baseline and after 6 and 12 months using the standard Medical Outcomes Study Short form( SF-36)questionnaire and the disease-specific Utility-Based Quality of life-Heart questionnaire(UBQ-H). | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Agewall, Professor, Principal Investigator — Oslo University Hospital. Department of Cardiology. Trondheimsveien 235, 0514 Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Trondheimsveien 235, Norway